CLINICAL TRIAL: NCT03581071
Title: Clinical Pharmacology Study of TS-143 in Nondialysis and Hemodialysis Patients with Chronic Kidney Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: TS143-01-02; JapicCTI-163383 (Other: JapicCTI)
Record Dates: First submitted 2018-04-18; First posted 2018-07-10 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2018-07

CONDITIONS: Chronic Kidney Disease
Keywords: Dialysis, CKD
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Step1:1mg in non-dialysis subject (Experimental)
  Interventions: Drug: TS-143
- Step2-1:1mg in hemodialysis subjects (Experimental)
  Interventions: Drug: TS-143
- Step2-2:6mg in non-dialysis subject (Experimental)
  Interventions: Drug: TS-143
- Step3-1:11㎎ in hemodialysis subjects (Experimental)
  Interventions: Drug: TS-143
- Step3-2:11㎎ in non-dialysis subject (Experimental)
  Interventions: Drug: TS-143

INTERVENTIONS:
Drug: TS-143

SUMMARY:
To evaluate the safety, pharmacokinetics, and pharmacodynamics in nondialysis (ND) and hemodialysis (HD) subjects with Chronic Kidney Disease (CKD) who receive a single administration of TS-143.

ELIGIBILITY:
Inclusion Criteria:

* Serum concentration of erythropoietin (EPO): <50 mIU/mL at screening test 1, 2, or 3
* Transferrin saturation ≥ 20% or ferritin ≥ 100 ng/mL at screening test 1
* Subjects meeting any of the following criteria

  1. Subjects who has not used erythropoiesis-stimulating agent (ESA) ≥ eight weeks from screening test 1
  2. Subjects who has used ESA, other than epoetin beta pegol, ≥ four weeks from screening test 1 and has met all of the following criteria A) to C).

A)The total ESA dosage for each week could be changed within a range of 50%, compared to the total ESA dosage for one week before screening test 1, for four weeks before screening test 1 B)Acceptable to discontinue ESA the day following screening test 1 to Follow-up 2 C)The fluctuating range of Hb concentration between screening tests 1 and 2 is within ±0.5 g/dL per week (the same criteria applied between screening test 2 and 3)

* Subjects who receive an explanation about the study before participating in the study and can understand the contents and are willing and able to provide written consent.

<Criteria for ND subjects>

* CKD subjects who never received dialysis and do not need to receive dialysis during the study period.
* Subjects with an Hb concentration at screening test 1 (ESA present at screening test 2) ≥ 10.0 g/dL to < 13.0 g/dL.
* Subjects with an eGFR at screening test 1 ≥ 15 mL/min/1.73m^2 to < 45 mL/min/1.73m^2.

<Criteria for HD subjects>

* Subjects who received hemodialysis (including diafiltration) three times per week ≥ 12 weeks from acquisition consent.
* Subjects with an Hb concentration at screening test 1 (ESA present at screening test 2) ≥ 10.0 g/dL to < 12.0 g/dL.

Exclusion Criteria:

* Subjects with anemia other than that caused by CKD.
* Subjects who have severe infection, systemic hematopathy (e.g. myelodysplastic syndrome, hemoglobinopathy), peptic ulcer or clear hemorrhagic lesion such as gastrointestinal hemorrhage
* Subjects with immune disorder with severe inflammation
* Subjects with uncontrolled secondary hyperparathyroidism
* Subjects who already had or will have a kidney transplantation
* Subjects who have a complication which requires treatment such as proliferative retinopathy, macular edema, or macular degeneration. Or, subjects who had a complication which required treatment such as proliferative retinopathy, macular edema, or macular degeneration within 12 months from screening test 1
* Subjects with congestive heart failure
* Subjects with a medical history of thrombotic disease in the six months from screening test 1
* Subjects with uncontrolled blood pressure; SBP > 170 mmHg or DBP > 100 mmHg at screening test 1 (ESA present, screening tests 1 and 2), (HD subject, evaluated before dialysis)

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2017-07-06 (Actual); Study Completion 2017-07-06 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | 8 days
  To evaluate the safety of TS-143 given single administration in CKD patients by incidence of adverse events which include abnormal electrocardiograms, vital signs, and clinical laboratory parameters.
Plasma concentrations of unchanged form (ng/mL) | 7 days
  The descriptive statistics (e.g., number of subjects, arithmetic mean, standard deviation) were calculated by dose group and evaluation timing.
Urinary excretions of unchanged form (ng/mL) | 24 hours
  The descriptive statistics (e.g., number of subjects, arithmetic mean, standard deviation) for the total urinary excretion (amount and fraction) were summarized by dose group.
Serum EPO concentration | 4 days
Reticulocyte count | 7 days
Plasma vascular endothelial growth factor (VEGF) concentration | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Okuyama, Study Director — Taisho Pharmaceutical Co., Ltd.
Locations (1):
- Taisho Pharmaceutical Co., Ltd selected site, Tokyo and Other Japanese City, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shinfuku A, Shimazaki T, Fujiwara M, Sato F, Watase H, Numazaki T, Kawakita Y, Mutoh M, Yamasaki H, Takayama N, Kato S, Sugimoto T, Maruyama J. Novel Compound Induces Erythropoietin Secretion through Liver Effects in Chronic Kidney Disease Patients and Healthy Volunteers. Am J Nephrol. 2018;48(3):157-164. doi: 10.1159/000492181. Epub 2018 Sep 3. PMID 30176654